CLINICAL TRIAL: NCT06093646
Title: Proposal to Address the Medium- to Long-term EBOLA Associated Psychological Distress and Psychosocial Problems in Mubende District in Central Uganda (Ebola+D Project)
Brief Title: Addressing Medium- to Long-term EBOLA Associated Psychological Distress and Psychosocial Problems in Central Uganda
Acronym: Ebola+D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: Ministry of Health, Uganda (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RGEK230305
Record Dates: First submitted 2023-08-07; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Ebola Virus Disease
Keywords: Ebola associated psychological distress
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Intervention Model Description: Screen participants attending 11 healthcare facilities at Mubende for psychological distress using the locally validated Luganda or English version of the WHO- Self Report Questionnaire (SRQ-20). Those individuals found to have significant psychological distress (a score of 6 and above) will be offered Ebola+D intervention. The intervention will include psycho-education, Problem Solving Therapy, antidepressant medication and referral to a supervising specialist mental health worker. A cohort of EVD affected individuals accessing the Ebola +D mental health intervention will be recruited and followed up for 12 months with assessments at three time points; baseline, 3 months and 12 months.
Masking Description: Masking will not be applied; eligible participants (with psychological distress) who consent to participate in this study will be offered the Ebola+D intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ebola+D intervention (Experimental): Ebola+D intervention will include psycho-education, Problem Solving Therapy, antidepressant medication and referral to a supervising specialist mental health worker.
  Interventions: Behavioral: Ebola+D intervention

INTERVENTIONS:
Behavioral: Ebola+D intervention — Ebola+D intervention will include psycho-education, Problem Solving Therapy, antidepressant medication and referral to a supervising specialist mental health worker.

SUMMARY:
Screen participants attending 11 healthcare facilities in Mubende District for psychological distress using the locally validated Luganda or English version of the WHO- Self Report Questionnaire (SRQ-20). Those individuals found to have significant psychological distress (a score of 6 and above) will be offered Ebola+D intervention [a stepped care collaborative delivery model to address the medium- to long-term EBOLA associated psychological Distress and psychosocial problems] . A cohort of Ebola Virus Disease (EVD) affected individuals accessing the Ebola +D mental health intervention will be recruited and followed up for 12 months with assessments at three time points; baseline, 3 months and 12 months.

DETAILED DESCRIPTION:
Ebola Virus Disease (EVD) is associated with high mortality, physical morbidity among patients and survivors, plus being associated with significant mental health and psychosocial problems among patients/survivors, their family members, members of the affected communities, health workers and volunteers. To support the medical services of Mubende district cope with the Ebola associated mental health and psychosocial problems, the Ministry of Health of Uganda has partnered with the MRC/UVRI & LSHTM Uganda Research Unit to implement a health systems strengthening project in the district entitled, 'Addressing the medium to long-term EBOLA associated psychological Distress and psychosocial problems in Mubende District in central Uganda (Ebola+D Project)'.

Methodology: The project will be undertaken in the 11 selected health care facilities in Mubende district. Members of the community attending these selected health care facilities will be screened for psychological distress using the locally validated Luganda or English version of the WHO- Self Report Questionnaire (SRQ-20). Those individuals found to have significant psychological distress (a score of 6 and above) will be offered Ebola+D intervention. A cohort of EVD affected individuals accessing the Ebola +D mental health intervention will be recruited and followed up for 12 months with assessments at three time points; baseline, 3 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Community member of Mubende district staying within the catchment area of the primary health care facility (PHCF);
* 18years and above,
* Able to communicate in either English or Luganda (local language spoken in the study region and the language into which the questionnaires will be translated),
* Has a WHO SRQ-20 score of 6 and above (except for Ebola survivors who are eligible even when their SRQ-20 score is either below or above 6). -

Exclusion Criteria:

* Unable to engage with the research process for any reason that may include sensory impairment or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Addressing the medium- to long-term EBOLA associated psychological Distress and psychosocial problems in Mubende District in central Uganda | Reduced psychological distress (SRQ-20 scores < 6) on two occasions ''4 weeks'' apart.
  Remission at ''3 months'' after completion of prescribed mental health treatment step(s) reduced psychological distress (SRQ-20 scores < 6) on two occasions ''4 weeks'' apart

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kinyanda, PhD, Principal Investigator — MRC/UVRI and LSHTM Uganda Research unit, Uganda
Locations (1):
- Mubende Regional Referal Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data collected from participants will be widely shared to support other research in the future, and may be shared anonymously with other researchers/authorities to effect policies /programs
Supporting Information: ICF, CSR
Time Frame: After the study (August 2024
Access Criteria: Data sets

REFERENCES:
- [Derived] Kyohangirwe L, Mpango RS, Tusiime C, Rutakumwa R, Ssebunnya J, Obuku A, Kiconco BE, Sekitoleko I, Sentongo H, Kalani K, Muhwezi W, Greco G, Baltra RA, Knizek BL, Kaleebu P, Mondelli V, Kyegombe N, Tenywa P, Amanyire P, Ssembajjwe W, Lund C, Kinyanda E. Protocol to develop and pilot a primary mental healthcare intervention model to address the medium- to long-term Ebola associated psychological distress and psychosocial problems in Mubende District in Central Uganda (the Ebola+D project). PLoS One. 2025 Aug 6;20(8):e0329591. doi: 10.1371/journal.pone.0329591. eCollection 2025. PMID 40768507